CLINICAL TRIAL: NCT01342861
Title: INAPEN Protocol for Impact of Breakfast Improvement on the Nutritional Status of Hospitalized Patients (INcidence de l'Amélioration du Petit-déjeuner Sur l'Etat Nutritinonel Des Patients hospitalisés)
Brief Title: INAPEN Protocol for Impact of Breakfast Improvement
Acronym: INAPEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Meaux (Other)
Responsible Party: Xavier Forceville, MD, PhD, CHdMeaux
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INAPEN
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Hospital Undernutrition; Malnutrition; Nutritional Deficiency
Keywords: protein supplementation; caloric intake; breakfast; transthyretin (prealbumin); albumin; Length of stay
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational period (Sham Comparator): A first period of follow-up on the 400 patients was designed to survey and evaluate current nutrition administration policy
  Interventions: Dietary Supplement: Addition of protein (milky food in the breakfast)
- Intervention period (Experimental): The second period of follow-up on the 400 patients was designed to evaluate the impacts of adding milky food to the breakfast and of educating health care professionals on the early detection of undernutrition.
  Interventions: Dietary Supplement: Addition of protein (milky food in the breakfast)

INTERVENTIONS:
Dietary Supplement: Addition of protein (milky food in the breakfast) — The main purpose of this study is to evaluate the efficacy of additional protein (adding milky food to the breakfast) in order to deliver an optimized protein and energy intake of 15.75 g and 559 Kcal, respectively.

SUMMARY:
Hospital undernutrition is a common health problem [1]. As a countermeasure, French hospitals have created a system of cross-function committees for feeding and nutrition called CLANs [Comité de Liaison pour l'alimentation et la nutrition] [2]. Potential actions for improving patient nutritional status include improving the characteristics of the food provided to increase both protein and calorie intake in at-risk patients that do not require enteral or parenteral nutrition. Looking at the various daily meals, the investigators considered that breakfast following the night fast would be the easiest meal to improve .

Condition Intervention Phase Patients scheduled for hospitalization of over 4 days Addition of protein (milky food in the breakfast) Current care

DETAILED DESCRIPTION:
INAPEN protocol for impact of breakfast improvement on the nutritional status of hospitalized patients (INcidence de l'Amélioration du Petit-déjeuner sur l'Etat Nutritinonel des patients hospitalisés)

Sponsored by Meaux Hospital (Centre Hospitalier de Meaux),

Financing: unrestricted grant from the French speaking society for enteral and parenteral nutrition [SFNEP: Société Francophone de nutrition entérale et parentérale].

Information provided by Meaux Hospital Center (Centre Hospitalier de Meaux) as per the protocol submitted to the SFNEP in 2009.

Purpose

Hospital undernutrition is a common health problem [1]. As a countermeasure, French hospitals have created a system of cross-function committees for feeding and nutrition called CLANs [Comité de Liaison pour l'alimentation et la nutrition] [2]. Potential actions for improving patient nutritional status include improving the characteristics of the food provided to increase both protein and calorie intake in at-risk patients that do not require enteral or parenteral nutrition. Looking at the various daily meals, we considered that breakfast following the night fast would be the easiest meal to improve .

Condition Intervention Phase Patients scheduled for hospitalization of over 4 days Addition of protein (milky food in the breakfast) Current care

Study Type: Interventional study in current care

Study design: Sequential cohorts, Efficacy study

Official title: Inapen Impact of breakfast improvement on the nutritional status of hospitalized patients (Incidence de l'amélioration du petit-déjeuner sur l'état nutritionnel des patients hospitalisés).

Further study details:

Primary outcome: Improvement of serum transthyretin (prealbumin) concentration changes between D0 to D7 Secondary outcomes: serum albumin concentration changes between D0 to D7, length of stay

Expected total enrollment: 800 patients (400 patients x 2).

Study start date: October 2009 Expected inclusion completion date: June 2011

Rationale:

It has long been known that more than half of hospitalized patients suffer from undernutrition [3-5]), consequently increasing length of stay of 2 to 6 days and morbidity [3]. Early nutrition has been shown to reduce length of stay and hospitalization costs [3, 6], but is mostly based on early enteral or parenteral nutrition. Our purpose was to evaluate the impact of an improved oral nutrition in mildly-challenged hospitalized patients. It is widely accepted that breakfast should deliver 25% of energy intake and nutritional requirements (ref4). A preliminary study found that the total protein and energy impact of breakfast in Meaux hospital was 4 g protein and 346 Kcal of total energy intake, whereas French institutional catering recommendations on nutrition (Groupe d'Etude des Marchés de Restauration Collective et de Nutrition, GEM RCN) stipulate 7.75 g of protein and 403 Kcal of energy.

The main purpose of this study is to evaluate the efficacy of additional protein (adding milky food to the breakfast) in order to deliver an optimized protein and energy intake of 15.75 g and 559 Kcal, respectively.

A first period of follow-up on the 400 patients was designed to survey and evaluate current nutrition administration policy. The second period of follow-up on the 400 patients was designed to evaluate the impacts of adding milky food to the breakfast and of educating health care professionals on the early detection of undernutrition. Efficacy will be evaluated based on increase in transthyretin concentrations, with special focus given to length of stay as a secondary end-point.

Eligibility Ages eligible for study: > 18 years. Both genders eligible for study.

Location and Contact Information France Rheumatology, Cardiology, Neurology, Pneumology departements Vascular and orthopedic surgery department

Study directorship and principal investigators Xavier Forceville, MD, PhD, Principal investigator Francois Thuillier, Pharmacist, CLAN chairman Karell Prieux-Lucas, Investigator Samia Touati, MD, Investigator

Further information

Study ID Number: CNIL : 909314 Health Authority: France CCTIRS : 09.358 (2009, september 10Th) Ethical committee: France, Ile-de-France XI (Saint Germain-en-Laye), August 17th, 2009

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for 8 days or more in the participant wards and capable of eating the proposed breakfast.

According to the current care procedure, patients receiving an information document and offered the possibility of refusal.

Exclusion Criteria:

* End of life defined as an absence of curative treatment (limitation of care)
* Enteral or parenteral nutrition
* Need for limitations on oral nutrition (i.e. post-surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
serum transthyretin (prealbumin) concentration | changes between D0 to D7 between the 2 cohorts
  Improvement of serum transthyretin (prealbumin) concentration changes between D0 to D7

SECONDARY OUTCOMES:
serum albumin concentration changes and length of stay | Changes between the 2 cohorts
  serum albumin concentration changes between D0 to D7, length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Meaux, Meaux, France

REFERENCES:
- [Background] Rapport complet de l'ANAES :Evaluation diagnostique de la dénutrition protéino-énergétique des adultes hospitalises. September 2003; http://www.has-sante.fr
- [Background] Reilly JJ Jr, Hull SF, Albert N, Waller A, Bringardener S. Economic impact of malnutrition: a model system for hospitalized patients. JPEN J Parenter Enteral Nutr. 1988 Jul-Aug;12(4):371-6. doi: 10.1177/0148607188012004371. PMID 3138447
- [Background] Circulaire DHOS/E1 N°2002-186 29/03/2002 relative à l'alimentation et la nutrition dans les établissements de santé: J off de la République Française 18/04/2002
- [Background] Kudsk KA, Tolley EA, DeWitt RC, Janu PG, Blackwell AP, Yeary S, King BK. Preoperative albumin and surgical site identify surgical risk for major postoperative complications. JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):1-9. doi: 10.1177/014860710302700101. PMID 12549591
- [Background] Edington J, Boorman J, Durrant ER, Perkins A, Giffin CV, James R, Thomson JM, Oldroyd JC, Smith JC, Torrance AD, Blackshaw V, Green S, Hill CJ, Berry C, McKenzie C, Vicca N, Ward JE, Coles SJ. Prevalence of malnutrition on admission to four hospitals in England. The Malnutrition Prevalence Group. Clin Nutr. 2000 Jun;19(3):191-5. doi: 10.1054/clnu.1999.0121. PMID 10895110
- [Background] Somanchi M, Tao X, Mullin GE. The facilitated early enteral and dietary management effectiveness trial in hospitalized patients with malnutrition. JPEN J Parenter Enteral Nutr. 2011 Mar;35(2):209-16. doi: 10.1177/0148607110392234. PMID 21378250